CLINICAL TRIAL: NCT07081412
Title: Home-Based Transcutaneous Remotely Monitored Posterior Tibial Neuromodulation System in Overactive Bladder: A Randomized Controlled Trial
Brief Title: Home-Based Transcutaneous Remotely Monitored Posterior Tibial Neuromodulation
Acronym: TRIP-HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Gokay Ozceltik, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRIP-HOME
Record Dates: First submitted 2025-07-12; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Overactive Bladder Syndrome; Overactive Bladder (OAB); Transcutaneous Posterior Tibial Nerve Stimulation (TTNS)
Keywords: overactive bladder; neuromodulation; Posterior Tibial Nerve Stimulation; Quality of Life
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Device (Experimental): T-PTNS treatment will be performed at home with an external generator and two surface electrode testers. Each T-PTNS session will consist of a test and treatment section. The treatment will be planned and carried out by the researchers.
  Treatment dose is 1 day/week, 30 minutes/session, totaling 12 sessions. Treatment Pulse Frequency: 20 Hz, Treatment Pulse Width: 200us (microsecond).
  Interventions: Device: Efficacy of remotely monitored transcutaneous posterior tibial nerve neuromodulation via a test device at 12 week and 12 month
- Sham Device (Placebo Comparator): These are devices that have the same physical appearance, interface and feedback features, but are prepared in a way that they will not provide electrical stimulation during the treatment session. They are delivered to the CRO by the project manager and are randomized through the CRO and given to the researchers with a code. The duration and frequency of treatment will be the same as the treatment group.
  Interventions: Device: Efficacy of remotely monitored transcutaneous posterior tibial nerve neuromodulation via a placebo device at 12 week

INTERVENTIONS:
Device: Efficacy of remotely monitored transcutaneous posterior tibial nerve neuromodulation via a test device at 12 week and 12 month — T-PTNS treatment will be performed at home with an external generator and two surface electrodes SmartUric medical device. Each T-PTNS session will consist of test and treatment sections. The treatment will be planned and carried out by researchers.
  The treatment dose is 1 day/week, 30 minutes/session, totaling 12 sessions. Treatment Pulse Frequency: 20 Hz, Treatment Pulse Width: 200us (microsecond).
  Arms: Test Device
Device: Efficacy of remotely monitored transcutaneous posterior tibial nerve neuromodulation via a placebo device at 12 week — These are devices that have the same physical appearance, interface and feedback features, but are prepared in a way that they will not provide electrical stimulation during the treatment session. They are delivered to the Contract Research Organization (CRO) by the project manager and are randomized through the CRO and given to the researchers with a code. The duration and frequency of treatment will be the same as the treatment group.
  Arms: Sham Device

SUMMARY:
To record the T-PTNS device (SmartUric) treatment performed by the patient at home via a mobile application in a remotely monitorable, secure and interactive manner with registration notes and a sham control group.

DETAILED DESCRIPTION:
1. Determination of candidate cases for the study
2. Conducting the eligibility assessment for the study according to the protocol (medical history, physical and urogynecological examination, USG, blood, urine analysis and/or culture tests if the researcher deems necessary)
3. Obtaining the informed consent form (VCF) from the cases who are found suitable and want to participate in the study
4. Creation of follow-up files specific to each patient in digital format and in hard copy for treatment follow-up.
5. Initial measurements will be made at the research center. The patient will be asked to fill out a three-day urinary diary, Overactive Bladder Assessment Form (OAB-V8) and International Incontinence Questionnaire-Short Form (ICIQ-UI-SF) for symptom and quality of life assessment. In addition, validated questionnaires such as Female Sexual Function Inventory-(FSFI) and Female Lower Urinary Tract Symptoms (ICIQ-FLUTS), Overactive Bladder Questionnaire-Short Form (OAB-q SF) given to the patient in hard copy will be used. These data will be taken as a starting point and recorded in the study follow-up files.
6. In order to provide and control T-PTNS usage training (The treatment will be applied by the patient at home), the researchers will provide training and sample application support to the patient until it is ensured that the patient can apply the treatment at home.
7. Start of 12-week T-PTNS treatment
8. The follow-up of treatment sessions can be monitored remotely by the researchers via the mobile application.
9. After the treatment session, the patient will be asked to complete the questionnaires included in the treatment follow-up (Three-day bladder diary, OAB-V8 and ICIQ-UI-SF) digitally from home via the mobile application.
10. The patients will be asked via phone in Weeks 2 or 3 which treatment group they think they are in and their answers will be recorded.
11. The patients who have completed their 12-session treatment will be invited to the hospital and will be asked to complete the Female Sexual Function Inventory (FSFI), Female Lower Urinary Tract Symptoms (ICIQ-FLUTS), Overactive Bladder Questionnaire-Short Form (OAB-q SF) forms given at the study center in addition to the surveys (OAB-V8, ICIQ-UI-SF, Three-day bladder diary) they completed via the mobile application.
12. According to the 12-week results;

    1. Patients whose treatment was completed with the real device and who benefited will be switched to maintenance treatment at the same treatment dose and once a month for 9 months.
    2. Patients who did not benefit in the sham treatment group will be given the real device and the same treatment procedure will be applied once a week, 30 minutes/session, for a total of 12 sessions. At the end of the 12 sessions, they will be called to the research center and the same evaluation procedure will be applied to the real device group. Patients who benefited in the sham group will be included in the 6-month maintenance treatment period. In the 3rd month maintenance treatment period, the interim evaluation will be made remotely via the mobile application.
13. Maintenance treatment will be monitored remotely in 3-month periods and the patients will fill out the digital questionnaires defined on the application every three months. The 3rd and 6th months will be repeated.
14. All patients who have completed their treatment will be called to the research center after one year of treatment and will be asked to complete the urinary diary and symptomatic questionnaire (OAB-V8 and ICIQ-UI_SF) evaluations as well as the Female Sexual Function Inventory-(FSFI), Female Lower Urinary Tract Symptoms (ICIQ-FLUTS), Overactive Bladder Questionnaire-Short Form (OAB-q SF) forms given in hard copy at the study center. At the same time, the researchers may call the patients who benefited after 12 sessions of sham treatment to the research center at the end of one year.
15. After all the evaluations, statistical analysis will be made at the end of the 12-week treatment and at the end of 1 year. In addition, if the researcher deems it appropriate, statistical analysis can be performed in the interim period (6 weeks, 3 months, 6 months).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥18 years old and female patients diagnosed with OAB* in Urology or Urogynecology outpatient clinics and who meet the inclusion criteria
2. Being able to continue their T-PTNS** treatment at home with the mobile application and accepting this,
3. Having a smartphone compatible with the application for T-PTNS and being able to use the application
4. Agreeing to be followed up for one year after treatment,
5. Having stopped all antimuscarinics for at least two weeks,
6. Being able to stand and use the toilet independently without difficulty,
7. Volunteers who are willing to participate, have been informed about the study and have given signed informed consent, stating that they can comply with the requirements and restrictions listed in the informed consent form (ICP) and this protocol.

Exclusion Criteria:

1. Patients under the age of 18
2. Patients who are pregnant according to the results of a pregnancy test with urine or blood test, or who are planning a pregnancy during the study period, or who are breastfeeding
3. Patients diagnosed with neurogenic bladder
4. Patients with Dabetes Mellitus whose blood sugar cannot be controlled
5. Patients with a history of allergic reactions on the skin
6. Cases with prolapse greater than Stage-2 according to the POP-Q staging system and extending beyond the hymen
7. Cases with a PVR evaluation of 100 ml and above with USG
8. Contraindications for T-PTNS treatment (patients with pacemakers, implantable defibrillators or metal prostheses
9. Patients with urinary tract infection*
10. Having had botox applied to the bladder or pelvic floor muscles within the last year
11. Having had a previous surgery related to the pelvic floor
12. Current TENS use in the pelvic region, back or legs
13. Having received PTNS treatment before
14. Use of Interstim or Bion
15. Those who do not accept the treatment or follow-up to be performed
16. Those who may have problems complying with the requirements of the study plan
17. Negative benefit/risk ratio determined by the investigator
18. Those who have been included in any other clinical trial or use of investigational drug/device therapy within 30 days before the study visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — born female
Enrollment: 50 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
3-Day Bladder Diary | Baseline, 12th week, and 12th month
  The 3-Day Bladder Diary is a structured patient-reported record used to evaluate urinary frequency, volume, fluid intake, urgency episodes, incontinence events, and nocturia across 3 consecutive days. Parameters recorded:
  * Time of each void
  * Voided volume (mL)
  * Fluid intake (time and volume)
  * Incontinence episodes (yes/no, with type if known)
  * Urgency (optional, often rated 0-3 or described qualitatively)
  * Nocturia episodes.
  At least 30% reduction in 24-hour urinary frequency or defined as at least a 50% reduction in the number of urgency sensations with or without incontinence and/or at least a 30% reduction in 24-hour urinary frequency via a urinary diary filled by the patient for three days.

SECONDARY OUTCOMES:
Overactive Bladder Questionnaire (OAB-V8) | Baseline, 12th week, and 12th month
  The Overactive Bladder Questionnaire (OAB-V8) is a validated screening tool used to identify the presence and severity of overactive bladder (OAB) symptoms. It includes 8 items that assess the bother associated with urgency, frequency, nocturia, and urge incontinence. Each item is rated on a Likert scale from 0 (not at all) to 5 (a very great deal), with a total score of ≥8 suggesting clinically relevant OAB. The OAB-V8 is commonly used in both clinical practice and research to support diagnosis and monitor symptom burden.
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | Baseline, 12th week, and 12th month
  The ICIQ-UI Short Form is a validated questionnaire used to assess the severity and impact of urinary incontinence on quality of life. It consists of four items evaluating the frequency, amount, and perceived interference of urinary leakage, as well as a self-diagnostic item for identifying incontinence type. The total score ranges from 0 to 21, with higher scores indicating greater severity.
The Overactive Bladder Quality of Life Short-Form (OAB-q SF) | Baseline, 12th week, and 12th month
  The OAB-q Short Form is a brief version of the original OAB-q designed to measure symptom bother and the quality of life impact in patients with overactive bladder. It is a patient-reported outcome measure used in clinical studies for efficient and reliable assessment of OAB-related impairments in daily functioning and well-being. The OAB-q Short Form consists of two main subscales:
  Symptom Bother Subscale (SB): Typically contains 6 items. Health-Related Quality of Life (HRQoL) Subscale: Typically contains 13 items. Each item is scored on a 6-point Likert scale (1-6).
  Scores are transformed to a 0-100 scale:
  Higher Symptom Bother scores indicate worse symptoms. Higher HRQoL scores indicate better quality of life. A 10-point change in the transformed score is generally considered clinically meaningful.
Female Sexual Function Index (FSFI) | Baseline, 12th week, and 12th month
  A 19-item questionnaire evaluating six domains of female sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. It is widely used in pelvic floor research and helps assess the broader quality-of-life effects of interventions. Scoring Range: 2-36 (higher scores = better function)
Female Lower Urinary Tract Symptoms Long Form Module (ICIQ-FLUTS Long Form) | Baseline, 12th week, and 12th month
  The ICIQ-FLUTS Long Form is a comprehensive questionnaire used to assess female lower urinary tract symptoms, including storage, voiding, and incontinence domains. Each item is scored from 0 to 4. It allows for detailed symptom characterization and is frequently utilized in clinical trials to evaluate the severity, bother, and treatment response in women with LUTS. Higher scores indicate greater symptom severity and greater bother.

CONTACTS AND LOCATIONS:
Overall Officials: Gokay Ozceltik, Associate Professor, Principal Investigator — Ege University, Faculty of Medicine, Department of Obstetrics and Gynaecology; Fuat Kızılay, Associate Professor, Study Chair — Ege University, Faculty of Medicine, Department of Urology; Sevtap Gunay Ucurum, Associate Professor, Study Chair — Izmir Katip Celebi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- EGE UNIVERSITY, FACULTY OF MEDICINE, Department of Obstetrics and Gynecology, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Ethical rules in scientific research protect the rights of participants and prevent the sharing of their personal data without their consent. In addition, commercial information may not be shared.

REFERENCES:
- [Background] • Cardozo, L., Rovner, E., Wagg, A., Wein, A., Abrams, P. 2023. Incontinence (7th Edition). Bristol UK: ICI-ICS. International Continence Society.